CLINICAL TRIAL: NCT02867995
Title: Efficacy of Glaucoma Drop Aids in Medication Compliance in the Patient Population at Boston Medical Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Manishi Desai, Faculty Sponsor, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-34905
Record Dates: First submitted 2016-08-07; First posted 2016-08-16 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Glaucoma
Keywords: glaucoma drop aid
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): No glaucoma drop aid control
- Eye Drop Aids (Active Comparator): Participants could be placed into one of the drop aid groups (Fabrication Autodrop Eye Drop Guide,Owen Mumford OP 6100 Autosqueeze, or the Simply Touch Eye Drop Applicator)
  Interventions: Device: Eye Drop Aid

INTERVENTIONS:
Device: Eye Drop Aid — Fabrication Autodrop Eye Drop Guide,Owen Mumford OP 6100 Autosqueeze, and the Simply Touch Eye Drop Applicator
  Arms: Eye Drop Aids

SUMMARY:
The purpose of this study is to determine whether glaucoma drop aids will be cost-effective in delivery of ophthalmic medications by improving medication compliance, visual function, and even decreasing medication waste in the patient population at Boston Medical Center (BMC).

DETAILED DESCRIPTION:
Patients being treated for their glaucoma at BMC's Yawkey Eye Clinic will be selected according to the inclusion and exclusion criteria. The three drop aids used in this study will be the Fabrication Autodrop Eye Drop Guide, Owen Mumford OP 6100 Autosqueeze, and the Simply Touch Eye Drop Applicator. Patients will be randomly placed on one of these drops aids for a total of 3 study groups or the no drop aid control, for a total of 4 groups. Prior to use of the drop aid, patients will be instructed on how to use the drop aid by a resident physician and a pre- intervention intraocular pressure check will be performed by the resident physician using an applicator. Intraocular pressure is the only adjustable risk factor for glaucoma; thus, glaucoma treatments slow progression of glaucoma by reducing intraocular pressure. In addition, patients will be requested to deliver their drops with the drop aid with every use. Furthermore, each patient will record the number of days taken to complete the glaucoma medication bottle while using the drop aid. At the 3 and 6 week marks, the patient will fill out a satisfaction survey. Patients will need to return to the clinic at the 6 week mark and can fill out the satisfaction survey at the clinic in addition to checking the intraocular pressure post-intervention. Thus, the number of subject contact will be two, pre and post-intervention, the duration of participation for each subject will be 6 weeks, and the patient will also be required to fill out two satisfaction surveys. The effectiveness of the drop aids will be compared to the two controls and measured with any changes in intraocular pressure readings, length of time to medication completion, and patient satisfaction according to the surveys.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or greater
* Currently on the same topical medication for treatment of glaucoma for a minimum of two months
* Patient of Boston University eye Associates
* Agrees to use the drop aid with each delivery, return to the clinic after 6 weeks of using the drop aid, document completion of medication drops and fill out survey at the end of the 6 weeks

Exclusion Criteria:

* Less than age 18 years
* Changes glaucoma medication within the past two month or recent glaucoma surgery
* Older than 89 years of age
* Not a patient of the Boston University eye associate

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manishi Desai, MD, Principal Investigator — Boston Medical Center; Haben Kefella, MD, Principal Investigator — Boston Medical Center; Avni Badami, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salyani A, Birt C. Evaluation of an eye drop guide to aid self-administration by patients experienced with topical use of glaucoma medication. Can J Ophthalmol. 2005 Apr;40(2):170-4. doi: 10.1016/S0008-4182(05)80028-6. PMID 16049530
- [Background] Ghate D, Edelhauser HF. Barriers to glaucoma drug delivery. J Glaucoma. 2008 Mar;17(2):147-56. doi: 10.1097/IJG.0b013e31814b990d. PMID 18344762
- [Background] Rivers PH. Compliance aids--do they work? Drugs Aging. 1992 Mar-Apr;2(2):103-11. doi: 10.2165/00002512-199202020-00004. PMID 1596593

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Eye Drop Aids
Started | 9 (Total patients consented) | 30 (Total patients consented)
Completed | 9 (Total patients completed) | 27 (Total patients completed)
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- No Drop Aid: No glaucoma drop aid received- control
- Drop Aid: Participants could be placed into one of the drop aid groups (Fabrication Autodrop Eye Drop Guide,Owen Mumford OP 6100 Autosqueeze, or the Simply Touch Eye Drop Applicator)
  Eye Drop Aid: Fabrication Autodrop Eye Drop Guide,Owen Mumford OP 6100 Autosqueeze, and the Simply Touch Eye Drop Applicator
- Total: Total of all reporting groups
Arm/Group | No Drop Aid | Drop Aid | Total
Number analyzed (Participants) | 9 | 30 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 17 | 19
  >=65 years | 7 | 13 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 16 | 18
  Male | 7 | 14 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 29 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 21 | 26
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 9 | 30 | 39
Glaucoma [Count of Participants; unit: Participants] | 9 | 30 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Intraocular Pressure Change
Description: Intraocular pressure (IOP) is measured by Goldman applanation in patients and is expressed in mmHg. The IOP, which is a routine check in the ophthalmic exam, was measured in the eye drop aid group prior to starting drop aid use and at six weeks while using drop aids. IOP was measured at baseline and at 6 weeks in the control group. A significant increase in IOP is defined as an increase of 4 mmHg or more, a significant decreases in IOP is defined as a decrease of 4mmHg or more. No significant change in the IOP is a change between 1-3 mmHg.
Time Frame: baseline and 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Eye Drop Aids
Number analyzed (Participants) | 9 | 27
Participants
  Significant increase in IOP | 0 | 4
  Significant decrease in IOP | 4 | 8
  No change in IOP | 5 | 15

2. Secondary Outcome: Number of Participants Stratified by the Number of Times Eye Was Missed When Inserting Eye Drops
Description: A question on the six week survey asked approximately how often the participant missed their eye when inserting eye drops. Response options included: missed inserting eye drops 0 times, missed inserting eye drops 1 time, missed inserting eye drops 2 times, or missed inserting eye drops 3 or more times.
Time Frame: 6 weeks
Population: Participants include those who were compliant with their drop aid device throughout the length of their medication bottle, as well as those who were non-compliant with their device group.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Eye Drop Aids
Number analyzed (Participants) | 9 | 27
Participants
  Missed inserting eye drops 0 times | 3 | 10
  Missed inserting eye drops 1 times | 5 | 8
  Missed inserting eye drops 2 times | 0 | 1
  Missed inserting eye drops 3 or more times | 1 | 2
  No Data Available | 0 | 6

3. Secondary Outcome: Satisfaction With Eye Drop Aid
Description: A question on the six week survey asked if the participant liked the eye drop aid. Response options included: liked the drop aid long term, did not like the drop aid, or did not use a drop aid. Results were stratified by the three drop aid types (Fabrication Autodrop Eye Drop Guide, Owen Mumford OP 6100 Autosqueeze, or the Simply Touch Eye Drop Applicator).
Time Frame: 6 weeks
Population: Participants include all enrolled patients who completed the study. The drop aid group was stratified into the three types of aids- AutoDrop, Autosqueeze, and Simply Touch.
Measure: Count of Participants; unit: Participants
Groups:
- AutoDrop: Patients placed in this group were given the Fabrication Autodrop Eye Drop Guide to instill their eye drops with
- Autosqueeze: Participants placed in this group were given the Owen Mumford OP 6100 Autosqueeze in order to instill their eye drops.
- Simply Touch: Participants placed in this group were given the Simply Touch Eye Drop Applicator in order to instill their eye drops.
Arm/Group | AutoDrop | Autosqueeze | Simply Touch | Control
Number analyzed (Participants) | 7 | 8 | 9 | 9
Participants
  Liked Drop Aid | 3 | 6 | 3 | 0
  Did Not Like Drop Aid | 4 | 2 | 4 | 0
  Did not use Drop Aid | 0 | 0 | 2 | 9

4. Secondary Outcome: Intent to Use Eye Drop Aid Long Term
Description: A question on the six week survey asked if the participant intended to use the eye drop aid long term. Response options included: would use the drop aid long term, would not use the drop aid long term, or did not use a drop aid. Results were stratified by the three drop aid types (Fabrication Autodrop Eye Drop Guide, Owen Mumford OP 6100 Autosqueeze, or the Simply Touch Eye Drop Applicator).
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | AutoDrop | Autosqueeze | Simply Touch | Control
Number analyzed (Participants) | 10 | 8 | 9 | 9
Participants
  Would use Drop Aid long term | 9 | 6 | 3 | 0
  Would not use Drop Aid long term | 1 | 2 | 4 | 0
  Did not use Drop Aid | 0 | 0 | 2 | 9

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Control: No glaucoma drop aid received- control
Arm/Group | Control | Eye Drop Aids
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/30
Other Adverse Events (participants affected / at risk) | 0/9 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT02867995/Prot_SAP_000.pdf